CLINICAL TRIAL: NCT02900586
Title: Understand the Behavior and the Knowledges of Patients Enrolled Into SIOUX Study
Brief Title: Behavior and Knowledges of Patients Enrolled Into SIOUX Study
Acronym: COM-Patient
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-01Obs-CHRMT
Record Dates: First submitted 2016-08-26; First posted 2016-09-14 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to contribute to the evaluation of SIOUX study by adding data about the choices of the observant patients, the mis-observant ones or the protocol deviations.

DETAILED DESCRIPTION:
The adherence to treatment for osteoporosis doesn't exceed 50% after one year. The SIOUX project about the inter-professional collaboration (attending physician with dispensary pharmacist) developed therapeutic patient education (TPE) plans and created follow-up booklets which were dealt to the patients who have to transmit it to their two medical professionals twice a year during three years one after one. The results after 18 months are encouraging about the improvement of adherence to treatment and about the lifestyle changes.

ELIGIBILITY:
Inclusion Criteria:

* patients enrolled into SIOUX study

Exclusion Criteria:

* cognitive troubles which prevent the patient to participate in individual interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoporotic patients who have been enrolled into SIOUX study
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Medication management | year 1
  semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Didier POIVRET, MD, Principal Investigator — CHR Metz-Thionville
Locations (1):
- Hôpital de Mercy - CHR Metz-Thionville, Metz, France

IPD SHARING:
Plan to Share IPD: No